CLINICAL TRIAL: NCT00254657
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Levetiracetam for Treatment of Pain Associated With Fibromyalgia
Brief Title: Levetiracetam for Treatment of Pain Associated With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: UCB Pharma (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: H5612-23162
Record Dates: First submitted 2005-11-15; First posted 2005-11-16 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Fibro; Keppra; Levetiracetam
MeSH Terms: conditions — Fibromyalgia | interventions — Levetiracetam

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Levetiracetam (Experimental)
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — Started with one 500 mg tablet/day and titrated upward as tolerated over 6 weeks by 500 mg/week to a maximum dose of 3000 mg/day.
  Other Names: Keppra
  Arms: Levetiracetam
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of levetiracetam in reducing the pain of fibromyalgia when compared to placebo. Levetiracetam, an anti-seizure drug, is currently FDA-approved and marketed for use in patients with seizures. Levetiracetam may relieve pain by reducing abnormal activity in the nervous system. A placebo is an inactive substance.

DETAILED DESCRIPTION:
The UCSF Pain Clinical Research Center (PCRC) will be conducting this investigator-initiated 9-week, randomized, double-blind, placebo-controlled, parallel group study of Levetiracetam. There will be a total of 6 study visits. Visit 1 is a screening visit to assess subject eligibility, followed by a one-week period of baseline daily pain and sleep assessments. Visit 2 (one week after Visit 1) subjects will be randomized in a 3/2-randomization scheme and administered study medication. Subjects randomized to the treatment group will start Levetiracetam at 1 tablet of 500/mg/day, and will titrate by 500mg each week to a maximum dose of 3000 mg/day. Visits 3, 4, 5, and 6 (occurring 2, 4, 6 and 8 weeks after started study drug) include safety and efficacy assessments. Study drug taper is initiated at Visit 6.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older.
2. Subjects must meet the 1990 American College of Rheumatology Criteria for the diagnosis of Fibromyalgia Syndrome.
3. Subjects at screening must have an average score of at least 40mm on the Visual Analog Scale (VAS) of the SF-McGill Pain Questionnaire; and at baseline must have an average score of at least 4/10 over the last 7 days on the Daily Pain Rating Scale.
4. Subjects must complete at least 4 diaries during the 7 days prior to randomization.
5. Subjects must discontinue use of steroids, muscle relaxants, anticonvulsants, sodium channel blockers, topical analgesics, and needle-based therapies, including trigger point injections and acupuncture, at least 1 week prior to starting study medication and agree to stay off such therapies throughout the study. Continuation of nonsteroidal anti-inflammatories, antidepressants and opiates are allowed, provided they have reached a stable dose prior to study entry and maintain a stable dose throughout the study.
6. Ability to understand and follow the instructions of the investigator, including completion of the study diaries as described in the protocol.
7. Ability to provide informed written consent.

Exclusion Criteria:

1. Subjects who have demonstrated a hypersensitivity to levetiracetam or who have been previously treated with it.
2. Subjects with severe liver or kidney insufficiency (AST, ALT, BUN, Creatinine more than twice the upper limit of the reference range).
3. Abnormal Westergen erythrocyte sedimentation rate (e.g. ESR >40 mm/min)
4. Abnormal antinuclear antibody (ANA≥1:160), or rheumatoid factor (RF>80 IU/ml)
5. Subjects with significant hematological disease, such as clotting disorders.
6. Subjects who have undergone trigger point injections or other needle-based therapies in the two weeks prior to dosing.
7. Subjects having other severe pain that may confound assessment of the pain due to the fibromyalgia.
8. Subjects taking or having taken any other experimental drugs, drugs not approved in the United States, or participating in or having participated in other clinical studies in the 2 months prior to this clinical trial.
9. Subjects who have a history of illicit drug or alcohol abuse within the last year.
10. Pregnant or lactating women.
11. Subjects who are considered unreliable as to medication compliance or adherence to scheduled appointments as determined by the investigators
12. Subjects who have serious or unstable medical or psychological conditions that in the opinion of the investigator(s), would compromise the subject's participation in the study.
13. Subjects involved in any unsettled litigation such as automobile accident, civil lawsuit, or worker's compensation pertaining to their fibromyalgia, current involvement in out-of-court settlements for litigation pertinent to their fibromyalgia, or are currently receiving monetary compensation as a result of any of the above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2004-03; Primary Completion 2005-03 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Weekly mean of average daily pain score as recorded in subjects' daily pain diaries and measured on an 11-point Likert scale with endpoints 0 ("no pain") and 10 ("worst pain") | Baseline to final week of treatment

SECONDARY OUTCOMES:
Sleep Interference over the past 24 hours as recorded in daily sleep diary on 11-point Likert scale (0 = "pain does not interfere with sleep" to 10 = "pain completely interferes with sleep" | Baseline to final week of treatment
  Change from mean score during baseline week to mean score during final week of treatment before tapering period began
Fibromyalgia Impact Questionnaire | Baseline to final week of treatment
  10-item, self-administered instrument designed to assess impact of fibromyalgia on physical functioning, work, fatigue, stiffness, anxiety and depression
Fibromyalgia Pain Now as measured using handheld 0-100 mm pain VAS (0 mm = "No pain" and 100 mm = "Worst pain imaginable" | Baseline to final week of treatment
Short-Form McGill Pain Questionnaire (SF-MPQ) | Baseline to final week of treatment
  Part 1: Fibromyalgia pain severity over past 7 days rate on 0-100 mm VAS; Part 2: Present pain intensity - 6 item category rating of pain "right now"; Part 3: Fifteen pain descriptors rated over past 7 days using 4 point intensity score (0= none to 3 = severe) and summed into sensory score and affective score
Fibromyalgia tender point score | Baseline to final week of treatment
  Number of days with headache in past 2 weeks reported (0=no headache; 1=1-2 days; 2=3-5 days; 3=6-9 days; 4=10-13 days; 5=headache all 14 days) and average headache severity rated on 0-10 NRS
Patient and Clinician Global Impression of Change | Final week of treatment
  Impression of change rated independently by subject and clinician on 1-7 category scale (1="very much improved", 2="much improved", 3="improved", 4="no change", 5="worse", 6="much worse", 7="very much worse"
Fibromyalgia tender point score | Baseline to end of treatment
  Manual Tender Point Survey with each site rated on 0-10 scale (0="no pain" and 10="worst pain imaginable"); "Fibromyalgia intensity score" represents mean sensitivity of 18 standardized tender point sites and "Control intensity score" represents mean sensitivity of 3 control sites

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Rowbotham, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States